CLINICAL TRIAL: NCT06639243
Title: Quick Yielding Modified Short-Distance Fenestration Technique for the Treatment of Complex Aortic Arch Diseases: a Multicenter Single-Arm Objective Performance Criteria Trial (QYM-Tech Study)
Brief Title: Quick Yielding Modified Short-Distance Fenestration Technique for the Treatment of Complex Aortic Arch Diseases: a Multicenter Single-Arm Objective Performance Criteria Trial(QYM-Tech Study)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Qingwei Ding, Medical Doctor, Sub-PI, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Qingwei Ding
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Thoracic Aortic Dissection; Thoracic Aortic Aneurysm (true Aneurysm); Thoracic Pseudoaneurysm; Penetrating Aortic Ulcer; Intramural Hematoma of the Thoracic Aorta
Keywords: Complex aortic arch diseases; Thoracic aortic dissection; Thoracic aortic aneurysm; Penetrating aortic ulcer; Quick Yielding Modified (QYM) technique
MeSH Terms: conditions — Dissection, Thoracic Aorta; Aortic Aneurysm, Thoracic; Penetrating Atherosclerotic Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- QTM Technique Treatment Arm (Experimental): In this study, all participants will undergo the Quick Yielding Modified (QYM) technique, which combines thoracic endovascular aortic repair (TEVAR) with in situ fenestration and revascularization of the supra-aortic branches. This technique is designed to treat patients with complex aortic arch diseases, including thoracic aortic dissection, true and pseudoaneurysms, penetrating aortic ulcers, and intramural hematomas. The procedure aims to provide a minimally invasive alternative to open surgery, allowing for the effective reconstruction of the aortic arch and its branches. The study will assess the safety and efficacy of this technique, with key outcomes including the incidence of major adverse events (MAE) and the long-term success of the treatment.
  Interventions: Device: QYM Technique

INTERVENTIONS:
Device: QYM Technique — The intervention in this study involves the application of the Quick Yielding Modified (QYM) technique for the treatment of complex aortic arch diseases. This procedure consists of two main components:
  1. Thoracic Endovascular Aortic Repair (TEVAR): This minimally invasive procedure utilizes a covered stent graft to exclude the diseased segment of the thoracic aorta, providing immediate protection against rupture and controlling blood flow.
  2. In Situ Fenestration and Revascularization of Supra-Aortic Branches: Following TEVAR, the QYM technique includes creating fenestrations in the stent graft to allow for the revascularization of the supra-aortic branches (such as the brachiocephalic, left common carotid, and left subclavian arteries). This is achieved through direct puncture and reconstruction of the branch vessels, ensuring adequate blood flow to these critical arteries while preserving their function.
  The combination of these techniques aims to achieve effective treatment out

SUMMARY:
Background: This study investigates the safety and efficacy of a novel surgical approach combining thoracic endovascular aortic repair (TEVAR) and in situ fenestration reconstruction of supra-aortic branches using the Quick Yielding Modified (QYM) technique. This procedure aims to address complex aortic arch diseases, providing an alternative to more invasive open surgical interventions.

Methods: This is a prospective, multicenter, single-arm, interventional study involving 87 patients across 3 centers. Eligible participants are adults aged 18-80 diagnosed with thoracic aortic dissection, thoracic aortic aneurysm (true or pseudo), penetrating aortic ulcer, or intramural hematoma, necessitating supra-aortic branch vessel reconstruction. The surgical protocol involves TEVAR combined with the QYM technique for fenestration and revascularization.

Primary Outcome: The primary endpoint is the incidence of major adverse events (MAE) within 30 days post-operation.

Secondary Outcomes: Secondary endpoints include 12-month aortic treatment success, all-cause mortality, aortic-related mortality, incidence of severe adverse events, occurrence of Type I/III endoleaks, stent graft migration, patency of revascularized branches, and rates of conversion to open surgery or reintervention due to aortic complications.

Inclusion/Exclusion Criteria: Key inclusion criteria include imaging-confirmed thoracic aortic disease requiring endovascular repair with a proximal landing zone in the aortic arch (Zone 0) and suitable anatomical features for stent placement. Patients with recent systemic infections, severe coronary artery involvement, or other significant comorbidities were excluded.

Follow-up and Statistical Analysis: Patients will undergo follow-ups at discharge, 30 days, 6 months, and 12 months post-surgery. Statistical analyses will include descriptive statistics of quantitative and categorical variables, with statistical significance set at a one-sided p-value < 0.025.

This study aims to provide critical insights into the clinical applicability of the QYM technique, potentially broadening therapeutic options for complex aortic arch diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Patients between 18 and 80 years of age.
2. Diagnosis: Patients with the following thoracic aortic conditions confirmed by imaging (CTA):

   * Thoracic aortic dissection
   * True thoracic aortic aneurysm
   * Thoracic pseudoaneurysm
   * Penetrating aortic ulcer
   * Intramural hematoma
3. Indication for Treatment: Patients requiring supra-aortic branch vessel reconstruction due to rupture, impending rupture, malperfusion syndrome, rapid expansion, uncontrolled pain, aneurysmal dilation, or for prophylactic reasons.
4. Proximal Landing Zone: Patients whose proximal stent landing zone is in Zone 0 of the aortic arch.
5. Aortic Anatomy:

   * Length of ascending aorta >4 cm (from the sinotubular junction to the proximal edge of the brachiocephalic artery).
   * Diameter of ascending aorta between 24 mm and 44 mm.
6. Access Vessel Anatomy:

   * Iliac artery diameter ≥7 mm.
   * Brachiocephalic artery diameter ≤24 mm, and length ≥20 mm.
7. Informed Consent: Patients who have been informed about the nature of the study and agreed to participate by signing the informed consent form.

Exclusion Criteria:

1. Infection: Patients with systemic infections within the last 3 months.
2. Recent Neck Surgery: Patients who underwent neck surgery within the past 3 months.
3. Coronary Involvement: Patients with disease extending to the coronary arteries or aortic valve.
4. Infectious or Autoimmune Diseases: Patients with conditions such as infectious aortic disease, large vessel vasculitis, or Marfan syndrome (or other connective tissue disorders).
5. Severe Vascular Conditions: Patients with severe stenosis, calcification, thrombosis, or tortuosity of the carotid or subclavian arteries.
6. Heart Transplant: Patients who have undergone heart transplantation.
7. Recent Cardiac Events: Patients who had a myocardial infarction or stroke within the last 3 months.
8. Advanced Heart Failure: Patients with New York Heart Association (NYHA) Class IV heart failure.
9. Active Gastrointestinal Conditions: Patients with active peptic ulcer disease or upper gastrointestinal bleeding within the past 3 months.
10. Hematologic Abnormalities:

    * Leukopenia (white blood cell count < 3×10⁹/L)
    * Acute anemia (hemoglobin < 90 g/L)
    * Thrombocytopenia (platelet count < 50×10⁹/L)
    * History of bleeding disorders or coagulopathy.
11. Renal Function: Patients with impaired renal function (creatinine > 265 µmol/L) or those with end-stage renal disease.
12. Pregnancy or Lactation: Pregnant or breastfeeding women.
13. Allergy to Contrast Media: Patients with an allergy to the contrast agents used in imaging.
14. Life Expectancy: Patients with an expected survival of less than 12 months.
15. Concurrent Research Participation: Patients involved in other drug or device trials.
16. Other Medical Conditions: Any other disease or condition that, in the opinion of the investigator, may interfere with the endovascular treatment or the patient's ability to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Major Adverse Events (MAE) Within 30 Days Post-Operation | 30 days post-operation
  This primary outcome measure evaluates the safety of the Quick Yielding Modified (QYM) technique by assessing the incidence of major adverse events (MAE) occurring within 30 days following the surgical intervention. Major adverse events include any significant complications that could impact patient health and recovery, such as stroke, myocardial infarction, aortic rupture, organ failure, or death. The goal is to determine the short-term safety profile of the intervention, providing critical information on its clinical viability for patients with complex aortic arch diseases. Data will be collected through patient monitoring, clinical assessments, and medical records during the specified follow-up period.

SECONDARY OUTCOMES:
Aortic Treatment Success Rate at 12 Months | Up to 12 months post-operation
  This secondary outcome measure assesses the effectiveness of the Quick Yielding Modified (QYM) technique by evaluating the rate of successful treatment of the aortic condition at 12 months post-intervention. Treatment success is defined as the absence of significant complications, such as re-intervention or aortic-related adverse events, and the proper functioning of the thoracic stent graft with no significant endoleaks. This measure provides insight into the long-term effectiveness and durability of the surgical intervention.
All-Cause Mortality | Up to 12 months post-operation
  This secondary outcome measure records the rate of all-cause mortality among participants within the study period, allowing for an evaluation of overall patient survival following the intervention. It provides crucial data on the safety and effectiveness of the QYM technique in comparison to the underlying risk of mortality associated with complex aortic arch diseases.
Aortic-Related Mortality | Up to 12 months post-operation
  This secondary outcome measure focuses specifically on mortality directly related to aortic conditions or complications arising from the surgical intervention. This measure helps to evaluate the long-term safety of the QYM technique concerning life-threatening aortic issues.
Incidence of Severe Adverse Events | Up to 12 months post-operation
  This measure tracks the occurrence of severe adverse events in participants, including complications such as stroke, myocardial infarction, and organ failure that are serious enough to require medical intervention. Monitoring these events provides a broader understanding of the risks associated with the procedure.
Occurrence of Type I or III Endoleaks | Up to 12 months post-operation
  This measure evaluates the incidence of Type I or Type III endoleaks following the intervention. Endoleaks are complications that can lead to re-intervention, and monitoring them is critical for assessing the effectiveness of the stent graft placement.
Rate of Stent Graft Migration | Up to 12 months post-operation
  This measure assesses the migration of the thoracic stent graft from its original position within the aorta. Stent migration can affect the success of the procedure and requires careful monitoring to ensure the stent remains securely in place.
Patency Rate of Revascularized Branch Vessels | Up to 12 months post-operation
  This measure evaluates the patency (openness and functionality) of the revascularized supra-aortic branches at follow-up visits. A high patency rate indicates successful reconstruction and blood flow restoration to these vessels.
Rate of Conversion to Open Surgery or Reintervention Due to Aortic Complications | Up to 12 months post-operation
  This measure tracks the incidence of participants who require conversion to open surgery or additional interventions due to complications related to the aorta after the initial procedure. It provides insight into the long-term risks and effectiveness of the QYM technique.
Incidence of Major Adverse Events (MAE) at 12 Months | 12 months post-operation
  This measure assesses the occurrence of major adverse events (MAE) within the 12-month follow-up period. Major adverse events include complications such as stroke, myocardial infarction, aortic rupture, or death. Monitoring the incidence of these events over the long term provides additional data on the safety and durability of the Quick Yielding Modified (QYM) technique.
Freedom from Aortic Rupture | 12 months post-operation
  This outcome tracks the percentage of participants who remain free from aortic rupture following the QYM technique over the course of 12 months. Aortic rupture is a life-threatening event, and the goal is to assess whether the intervention effectively prevents this complication in patients with complex aortic arch diseases.
Freedom from Reintervention | 12 months post-operation
  This measure evaluates the percentage of participants who do not require additional surgical or endovascular interventions on the thoracic aorta or supra-aortic branches after the initial procedure. The goal is to assess the long-term effectiveness of the QYM technique and its ability to prevent the need for further treatments.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Vascular Surgery, General Surgery Clinical Center, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China., Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shu C, Fan B, Luo M, Li Q, Fang K, Li M, Li X, He H, Wang T, Yang C, Xue Y, Gao H, Zhao J. Endovascular treatment for aortic arch pathologies: chimney, on-the-table fenestration, and in-situ fenestration techniques. J Thorac Dis. 2020 Apr;12(4):1437-1448. doi: 10.21037/jtd.2020.03.10. PMID 32395281
- [Background] Matsuda H, Fukuda T, Iritani O, Nakazawa T, Tanaka H, Sasaki H, Minatoya K, Ogino H. Spinal cord injury is not negligible after TEVAR for lower descending aorta. Eur J Vasc Endovasc Surg. 2010 Feb;39(2):179-86. doi: 10.1016/j.ejvs.2009.11.014. Epub 2009 Dec 3. PMID 19962330
- [Background] Wang J, Jin T, Chen B, Pan Y, Shao C. Systematic review and meta-analysis of current evidence in endograft therapy vs medical treatment for uncomplicated type B aortic dissection. J Vasc Surg. 2022 Oct;76(4):1099-1108.e3. doi: 10.1016/j.jvs.2022.03.876. Epub 2022 Apr 4. PMID 35390485